CLINICAL TRIAL: NCT07028047
Title: Evaluation for Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Anti-tumor Activity of WGc-043 Injection in Patients With Advanced Malignant Solid Tumors: Phase I Study
Brief Title: Evaluation of WGc-043 Injection in Advanced Solid Tumors: Phase I Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Assistant Dean and Director of Nasopharyngeal Department, Sun Yat-sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WGc-043-002
Record Dates: First submitted 2025-06-09; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Advanced EBV-positive Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WGc-043 Injection, Dose 1 (Experimental)
  Interventions: Biological: WGc-043 Injection
- WGc-043 Injection, Dose 2 (Experimental)
  Interventions: Biological: WGc-043 Injection
- WGc-043 Injection, Dose 3 (Experimental)
  Interventions: Biological: WGc-043 Injection
- WGc-043 Injection, Dose 4 (Experimental)
  Interventions: Biological: WGc-043 Injection
- WGc-043 Injection, Extended dosage (Experimental)
  Interventions: Biological: WGc-043 Injection

INTERVENTIONS:
Biological: WGc-043 Injection — WGc-043 Injection, intramuscular injection

SUMMARY:
Epstein-Barr virus (EBV) is an important tumor-associated virus. In 1997, the World Health Organization (WHO) officially classified EBV as a Group 1 carcinogen, as it is implicated in the pathogenesis of various epithelial malignancies and multiple types of lymphomas. Epithelial malignancies associated with EBV infection include nasopharyngeal carcinoma, gastric cancer, colorectal cancer, breast cancer, cervical cancer, prostate cancer, and oral cancer, among others. Currently, optimal therapeutic strategies for EBV-associated solid tumors remain lacking, particularly in patients with recurrent, metastatic, or refractory disease. Furthermore, although EBV infection plays a significant role in the development and progression of EBV-positive tumors and may influence patient prognosis, there are currently no precision therapeutic approaches specifically targeting EBV-positive lymphomas. Thus, treatment options for this patient population warrant further attention.

WGc-043 injection is a therapeutic tumor vaccine based on messenger RNA (mRNA) targeting tumor-specific antigens expressed in EBV-positive tumors. This Phase I clinical trial aims to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, and preliminary antitumor activity of WGc-043 in patients with advanced EBV-positive malignant solid tumors, thereby providing a scientific basis for subsequent clinical development.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years at the time of screening;
2. Histologically or cytologically confirmed locally recurrent or metastatic EBV-positive solid tumors that are not amenable to curative treatment;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
4. Estimated life expectancy of ≥3 months;
5. At least one measurable lesion; previously irradiated lesions cannot be considered as target lesions unless there is evidence of significant progression;
6. Adequate major organ function, with organ function parameters meeting the criteria specified in the protocol;
7. Women of childbearing potential (WOCBP) or male subjects must have no plans for pregnancy during the study and must agree to use effective contraception (including one or more non-pharmacologic contraceptive methods or complete abstinence from heterosexual intercourse) or safety measures during the trial and for 6 months after discontinuation of treatment;
8. Ability to understand and voluntarily sign the written informed consent form prior to participation in the trial;
9. Ability to communicate effectively with the investigator and comply with the protocol requirements throughout the trial.

Exclusion Criteria:

1. Patients with a history of other malignancies, except for those with a history of skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix, gastrointestinal mucosal carcinoma, or other malignancies deemed by the investigator to be eligible for inclusion, provided that these cancers have been cured and have not recurred within 5 years prior to screening.
2. Patients with symptomatic central nervous system (CNS) metastases or leptomeningeal metastases, or those with evidence indicating that CNS or leptomeningeal metastases are not well-controlled, as judged by the investigator to be unsuitable for inclusion.
3. Patients with known uncontrolled cardiac symptoms or diseases, such as: New York Heart Association (NYHA) Class II or higher heart failure, unstable angina, myocardial infarction within the past 6 months, or clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
4. Any active autoimmune disease or a history of autoimmune disease.
5. Any uncontrolled clinical condition or other major medical illness that, in the judgment of the investigator, may interfere with the ability to provide informed consent, confound the interpretation of trial results, pose a risk to the patient's participation in the trial, or otherwise affect the achievement of trial objectives-including, but not limited to, uncontrolled pleural effusion, pericardial effusion, or ascites as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | During one year after initial treatment
Safety: Type, frequency, and severity of treatment-related adverse events as assessed by CTCAE V5.0 | During one year after initial treatment
MTD/RP2D | During one year after initial treatment

SECONDARY OUTCOMES:
Preliminary antitumor activity: Objective response rate (ORR) | During one year after initial treatment
Preliminary antitumor activity: Disease control rate (DCR) | During one year after initial treatment
Preliminary antitumor activity: Duration of response (DoR) | During one year after initial treatment
Preliminary antitumor activity: Progression-free survival (PFS) | During one year after initial treatment
Preliminary antitumor activity: 1-year survival rate | During one year after initial treatment
Immunogenicity: The level of antigen-specific T cells | During one year after initial treatment
Pharmacokinetics (PK) characteristics: Maximum Plasma Concentration [Cmax] of mRNA | During one year after initial treatment
Pharmacokinetics (PK) characteristics: Maximum Plasma Concentration [Cmax] of cationic lipids | During one year after initial treatment